CLINICAL TRIAL: NCT00930956
Title: Resistant Starch Type 2 and Cross Linked Resistant Starch Type 4 on Blood Glucose
Brief Title: Comparison of Different Types of Resistant Starch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Mark Haub, Kansas State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KSUHML09-RS
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2009-06

CONDITIONS: Postprandial Hyperglycemia
Keywords: Diabetes; Obesity; Hyperglycemia; Dietary Fiber; Wheat; Grain
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Obesity | interventions — Resistant Starch; high-amylose maize type 2 resistant starch, maize

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dextrose (Active Comparator): 30 g of carbohydrate via Sun-Dex OGTT beverage
  Interventions: Dietary Supplement: Resistant Starch
- RS Type 2 (Experimental): 30g Resistant Starch Type 2 (Hi-Maize 260, National Starch)
  Interventions: Dietary Supplement: Resistant Starch
- RS Type 4 (cross linked) (Experimental): 30g of cross linked RS type 4 (Fibersym RW, MGP Ingredients, Inc.)
  Interventions: Dietary Supplement: Resistant Starch

INTERVENTIONS:
Dietary Supplement: Resistant Starch — 30 g of carbohydrate per Arm
  Other Names: Hi-Maize 260; Fibersym RW

SUMMARY:
This study is to determine whether different types of resistant starch have different effects on blood glucose in healthy adults.

DETAILED DESCRIPTION:
Each volunteer will visit the laboratory in a 10-12 hour fasted state on three occasions over a three-week period, up to two visits/wk, with at least 48 hours between visits. Volunteers will be asked to refrain from vigorous physical activity and the consumption of alcohol the day before each testing visit. Randomization using a Latin Square design was applied to minimize confounding issues associated with the order of administration.

In the morning of each test, a finger-prick capillary blood samples will be collected to determine fasting (baseline) blood glucose levels. The volunteers will then consume the test solution assigned for that trial. Ten minutes will be allowed for the test solution to be consumed. Over the two hours following the start of each test, finger-prick capillary blood samples were collected at 30, 60, 90, and 120 min. Blood glucose levels will be immediately measured in duplicate using an automated blood glucose analyzer (YSI 2300, Yellow Springs, OH). Analysis of the collected sample was repeated if the difference between duplicate samples was greater than 0.1 mmol/L. Once the samples were analyzed, the data was entered and the incremental area under the curve was calculated using the trapezoidal model (GraphPad v5.0, La Jolla, CA).

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy

Exclusion Criteria:

* diagnosis of any chronic disease
* wheat allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Acute response -- fasting and 30, 60, 90 and 120 minutes post-ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Haub, Ph.D., Principal Investigator — Kansas State University
Locations (1):
- Human Metabolism Laboratory (K-State Univ.), Manhattan, Kansas, United States